CLINICAL TRIAL: NCT02796651
Title: A Randomized, Double-blind, Placebo-controlled, Incomplete Unbalanced, Crossover Study to Assess the Efficacy and Safety of Three Doses of Formoterol Fumarate in Pressair® Compared With Perforomist® Inhalation Solution (20 and 40 μg Open-label) in Moderate to Severe COPD Patients With Reversible Airway Disease.
Brief Title: Formoterol Dose Ranging Study (ACHIEVE Duaklir USA Phase IIb)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D6571C00002
Record Dates: First submitted 2016-06-07; First posted 2016-06-13 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Chronic Obstructive Pulmonary Disease - COPD
Keywords: Perforomist; Pressair; COPD; Cigarette smoking; Formoterol fumarate; long-acting β2-adrenergic agonists (LABA); long-acting muscarinic antagonists (LAMA)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cigarette Smoking | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Formoterol 6 μg (Experimental): Participants received formoterol fumarate 6 μg administered via Pressair twice daily (BID).
  Interventions: Drug: Formoterol fumarate (6 μg)
- Formoterol 12 μg (Experimental): Participants received formoterol fumarate 12 μg administered via Pressair BID.
  Interventions: Drug: Formoterol fumarate (12 μg)
- Formoterol 24 μg (Experimental): Participants received formoterol fumarate 24 μg administered via Pressair BID.
  Interventions: Drug: Formoterol fumarate (12 μg)
- Placebo (Placebo Comparator): Participants received placebo to formoterol fumarate administered via Pressair BID.
  Interventions: Drug: Placebo for formoterol fumarate
- Formoterol 20 μg (Experimental): Participants received Perforomist inhalation solution and were instructed to take one puff from each of the two Pressair inhalers or to inhale one vial from the Perforomist 20 μg inhalation solution BID for 7 ± 1 consecutive days.
  Interventions: Drug: Formoterol furmarate (20 μg)
- Formoterol 40 μg (Experimental): Participants received Perforomist 40 μg (2 vials of Performist 20 μg) as a single dose of administration.
  Interventions: Drug: Formoterol fumarate (40 μg)

INTERVENTIONS:
Drug: Formoterol fumarate (6 μg) — Oral Inhalation (by Pressair® Dry Powder Inhaler, DPI)
  Other Names: Formoterol (Pressair®)
  Arms: Formoterol 6 μg
Drug: Formoterol furmarate (20 μg) — Oral Inhalation (via a standard jet nebulizer connected to an air compressor.
  Other Names: Perforomist® Inhalation Solution
  Arms: Formoterol 20 μg
Drug: Placebo for formoterol fumarate — Oral Inhalation (by Pressair® Dry Powder Inhaler, DPI)
  Other Names: Placebo (Pressair®)
  Arms: Placebo
Drug: Formoterol fumarate (12 μg) — Oral Inhalation (by Pressair® Dry Powder Inhaler, DPI)
  Other Names: Formoterol (Pressair®)
  Arms: Formoterol 12 μg; Formoterol 24 μg
Drug: Formoterol fumarate (40 μg) — Oral Inhalation (via a standard jet nebulizer connected to an air compressor.
  Other Names: Perforomist® Inhalation Solution
  Arms: Formoterol 40 μg

SUMMARY:
To assess the bronchodilation of three doses of formoterol fumarate (6 μg, 12 μg and 24 μg) twice daily (BID) administered via Pressair® compared to placebo and to open-label nebulized formoterol fumarate (20 μg and 40 μg).

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, 5-period incomplete unbalanced crossover, placebo and active comparator (open-label) controlled, multicenter clinical trial to assess the efficacy and safety of three doses of formoterol fumarate (6 μg, 12 μg and 24 μg) BID administered via Pressair® compared to placebo and to open-label formoterol fumarate (20 μg BID and 40 μg single dose) administered as an inhalation solution via a standard jet nebulizer (with a mouthpiece) connected to an air compressor (Perforomist® Inhalation Solution). The drug product is an inhalation powder comprising of micronized aclidinium bromide and micronized formoterol fumarate with α-lactose monohydrate as the carrier, presented in a breathactuated device-metered dry-powder inhaler (DPI). It has been approved under the trademarks of Genuair® and/or Pressair® in some territories.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or non-pregnant, non-lactating female patients aged ≥40.
* Patients with a diagnosis of COPD (GOLD guidelines, 2016) for a period of at least 6 months prior to Visit 1.
* Patients with moderate to severe stable COPD: post-bronchodilator FEV1 ≥ 30% and <80% of the predicted normal and post-bronchodilator FEV1/FVC < 70% at Visit 1.
* Patients with reversible airway obstruction defined as an increase in FEV1 of at least 12% and 200 mL over the baseline value after four inhalations of albuterol sulfate 108 µg via a pMDI at Visit 1.
* Current or former-smokers, with a smoking history of ≥ 10 pack-years.
* Patients able to perform acceptable and repeatable pulmonary function testing for FEV1 according to the American Thoracic Society (ATS)/European Respiratory Society (ERS) 2005 criteria at Visit 1.
* Patients eligible and able to participate in the study and who had signed an Informed Consent Form prior to initiation of any study-related procedures.

Exclusion Criteria:

* Patients with asthma.
* Any respiratory tract infection (including the upper respiratory tract) or COPD exacerbation (including the mild COPD exacerbation) within 6 weeks prior to Visit 1 or during the run-in period.
* Patients hospitalized for a COPD exacerbation (an emergency room visit for longer than 24 hours is considered a hospitalization) within 3 months prior to Visit 1.
* Clinically significant respiratory conditions other than COPD.
* Patients who in the investigator's opinion may need to start a pulmonary rehabilitation program during the study and/or patients who started/finished it within 3 months prior to Visit 1.
* Use of long-term oxygen therapy (≥ 15 hours/day).
* Patients who do not maintain regular day/night, waking/sleeping cycles including night shift workers.
* Clinically significant cardiovascular conditions.
* Patients with uncontrolled Type I or Type II diabetes, uncontrolled hypo-or hyperthyroidism, hypokalaemia, or hyperadrenergic state, uncontrolled hypertension.
* Patients with history of long QT syndrome or whose QTc (calculated according to Fridericia's Formula QTc=QT/RR1/3) > 470 ms as indicated in the centralized reading report assessed at Visit 1.
* Patients with clinically significant abnormalities in the laboratory tests, ECG parameters (other than QTc) or in the physical examination at Visit 1 that might compromise patient safety.
* Patients with a history of hypersensitivity reaction to an inhaled medication or any component thereof, including paradoxical bronchospasm.
* Patients with known narrow-angle glaucoma, symptomatic bladder neck obstruction, acute urinary retention or symptomatic unstable prostate hypertrophy.
* History of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years other than basal or squamous cell skin cancer.
* Patients with any other serious or uncontrolled physical or mental dysfunction.
* Patients with a history (within 2 years prior to screening) of drug and/or alcohol abuse that may prevent study compliance based on the Investigator judgment.
* Patients unlikely to be cooperative or who cannot comply with the study procedures.
* Patients treated with any investigational drug within 30 days (or 6 half-lives, whichever is longer) prior to Visit 1.
* Patients who intended to use any concomitant medication not permitted by this protocol or who had not undergone the required washout period for a particular prohibited medication.
* Patients unable to give consent, or patients of consenting age but under guardianship, or vulnerable patients.
* Any other conditions that, in the investigator's opinion, might render the patient to be unsuitable for the study.
* Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff and/or site staff), or patients employed by or relatives of the employees of the site or sponsor.
* Previous randomization in the present study D6571C00002.

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2016-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H. Gotfried, MD, Principal Investigator — 1112 East McDowell Road, Phoenix, AZ 85006, United States.
Locations (20):
- United States (20):
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Celebration, Florida
  - Research Site, Clearwater, Florida
  - Research Site, DeLand, Florida
  - Research Site, Orlando, Florida
  - Research Site, Lawrenceville, Georgia
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Charlotte, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Easley, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Rock Hill, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Boerne, Texas
  - Research Site, Killeen, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was carried on 132 participants with moderate to severe chronic obstructive pulmonary disease (COPD) & reversible airway disease in the United States of America (USA; 21 sites) & were randomized to one of treatment sequences (each with 5 periods of different treatment, separated by wash-out period of 7 (+/1) days after treatment period).
Pre-assignment Details: After signature of the informed consent, participants who were taking prohibited medication performed a wash-out period and were given Atrovent (2 puffs 4 times/day) before Screening and during the run-in period. All participants were provided with rescue drug (albuterol) and Atrovent to be taken during the wash-out between treatment periods.
Groups:
- Total Participants: All patients were randomized in a treatment sequence containing 5 treatment periods. All patients received FF12 and Perforomist 20 mcg, 90% received FF6, FF24 and Perforomist 40 mcg, and only 30% received placebo. Treatment was double blind for FF in Pressair, and open label for Perforomist. If treatment was FF6, FF12, FF24 or placebo, patients received two identical Pressair dry powder inhalers (DPI) and were instructed to take 1 puff from each of the inhalers in the morning and in the evening for 7 days. If treatment was Perforomist 20 mcg, patients were instructed to take 1 vial in the morning and 1 vial in the evening for 7 days. Treatment with Perforomist 40 mcg was a single dose administration.
  Note: 132 participants were randomized. But, one participant was excluded from the ITT analysis set as the participant did not have a post-baseline forced expiratory volume in 1 second (FEV1) measurement.
Period: Overall Study
Arm/Group | Total Participants
Started | 132
Formoterol Fumarate (FF) 6 μg (Participants had 1 puff each from 2 identical Pressair DPI (FF 6μg & placebo) in morning & evening) | 107
Formoterol Fumarate (FF) 12 μg (Participants had 1 puff each from 2 identical Pressair DPI (FF 12μg & placebo) in morning & evening) | 121
Formoterol Fumarate (FF) 24 μg (Participants had 1 puff each from 2 identical Pressair DPI (FF 24μg & placebo) in morning & evening) | 105
Perforomist 20 μg (Participants took 1 vial of Perforomist 20μg oral nebulization solution in morning & evening) | 118
Perforomist 40 μg (Participants took 1 dose of 2 vials of Perforomist 20μg oral nebulization solution on Day 1 morning) | 108
Placebo (Lactose Monohydrate) (Participants had 1 puff from Pressair DPI (FF 6/12/24 μg matching placebo) in morning & evening) | 38
Completed | 106
Not Completed | 26
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 4
Not completed — Lack of Efficacy | 1
Not completed — Other | 10

BASELINE CHARACTERISTICS:
Population: The ITT analysis set: Consisted of all randomized participants who received at least 1 dose of investigational product (IP) and had a baseline FEV1 value and at least 1 post-baseline FEV1 measurement, regardless of a participant's adherence to the randomized treatment.
Groups:
- Overall Study Total: All patients were randomized in a treatment sequence containing 5 treatment periods. All patients received FF12 and Perforomist 20 mcg, 90% received FF6, FF24 and Perforomist 40 mcg, and only 30% received placebo. Treatment was double blind for FF in Pressair, and open label for Perforomist. If treatment was FF6, FF12, FF24 or placebo, patients received two identical Pressair DPI and were instructed to take 1 puff from each of the inhalers in the morning and in the evening for 7 days. If treatment was Perforomist 20 mcg, patients were instructed to take 1 vial in the morning and 1 vial in the evening for 7 days. Treatment with Perforomist 40 mcg was a single dose administration.
  Note: 132 participants were randomized. But, one participant was excluded from the ITT analysis set as the participant did not have a post-baseline forced expiratory volume in 1 second (FEV1) measurement.
Arm/Group | Overall Study Total
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (7.5)
Age, Customized [Number; unit: Participants]
  <50 years | 5
  ≥50 to <65 years | 78
  ≥65 years | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 65

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Normalized Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve (AUC) Over the 12 h Period Immediately After Morning Study Drug Administration, AUC0-12/12h at Day 7 on Treatment
Description: To assess the bronchodilation of 3 doses of formoterol fumarate (6 μg, 12 μg and 24 μg) twice daily (BID administered via Pressair® compared to placebo and to open-label nebulised formoterol fumarate(20 μg).
  Pre-dose spirometry was performed before the morning daily dose at Day 1 and Day 7 of each treatment period. Two sets of measurements were performed during the hour preceding the scheduled morning study drug administration, allowing approximately 30 minutes between them.
  Note: Perforomist® 40 μg treatment periods lasted for 1 day only. Hence, was not included in the calculation.
Time Frame: Day 7: 30 min, 1 to 4 hours, 6 hours, 9 hours and 12 hours post-dose
Population: The ITT analysis set consisted of all randomized participants who received at least 1 dose of investigational product (IP) and had a baseline FEV1 value and at least 1 post-baseline FEV1 measurement, regardless of a participant's adherence to the randomized treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Litre/Hour
Groups:
- Formoterol Fumarate 6 μg: Randomized participants received 2 puffs of Formoterol Fumarate 6 μg oral inhalation powder using Pressair® dry powder inhaler (DPI) in the morning and evening for 7 (±1) days
- Formoterol Fumarate (FF) 12 μg: Randomized participants received two identical Pressair dry powder inhaler (DPI; FF 12 μg and placebo) and were instructed to take one puff from each of the two Pressair DPI in the morning and in the evening for 7 days
- Formoterol Fumarate (FF) 24 μg: Randomized participants received two identical Pressair dry powder inhaler (DPI; FF 24 μg and placebo) and were instructed to take one puff from each of the two Pressair DPI in the morning and in the evening for 7 days
- Perforomist 20 μg: Randomized participants received 1 vial of Perforomist 20 μg oral nebulization solution via a jet nebulizer in the morning and evening for 7 (±1) days
- Placebo (Lactose Monohydrate): Randomized participants received two identical Pressair dry powder inhaler (DPI; FF 6/12/24 μg and placebo) and were instructed to take one puff from each of the two Pressair DPI in the morning and in the evening for 7 days
Arm/Group | Formoterol Fumarate 6 μg | Formoterol Fumarate (FF) 12 μg | Formoterol Fumarate (FF) 24 μg | Perforomist 20 μg | Placebo (Lactose Monohydrate)
Number analyzed (Participants) | 105 | 118 | 104 | 116 | 35
Litre/Hour | 0.108 [0.073 to 0.143] | 0.117 [0.082 to 0.151] | 0.161 [0.125 to 0.197] | 0.122 [0.087 to 0.156] | 0.000 [-0.055 to 0.054]
Statistical Analysis 1: Comparison: Formoterol Fumarate 6 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.108, 95% CI 2-sided [0.055 to 0.161]
Statistical Analysis 2: Comparison: Formoterol Fumarate (FF) 12 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.117, 95% CI 2-sided [0.064 to 0.171]
Statistical Analysis 3: Comparison: Formoterol Fumarate (FF) 24 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.162, 95% CI 2-sided [0.107 to 0.216]
Statistical Analysis 4: Comparison: Perforomist 20 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.122, 95% CI 2-sided [0.069 to 0.175]
Statistical Analysis 5: Comparison: Formoterol Fumarate 6 μg vs Formoterol Fumarate (FF) 12 μg; Test type: Superiority; p = 0.556, Mixed Models Analysis; LSMean difference = 0.009, 95% CI 2-sided [-0.021 to 0.039]
Statistical Analysis 6: Comparison: Formoterol Fumarate 6 μg vs Formoterol Fumarate (FF) 24 μg; Test type: Superiority; p = 0.001, Mixed Models Analysis; LSMean difference = 0.053, 95% CI 2-sided [0.021 to 0.085]
Statistical Analysis 7: Comparison: Formoterol Fumarate 6 μg vs Perforomist 20 μg; Test type: Superiority; p = 0.365, Mixed Models Analysis; LSMean difference = 0.014, 95% CI 2-sided [-0.016 to 0.044]
Statistical Analysis 8: Comparison: Formoterol Fumarate (FF) 12 μg vs Formoterol Fumarate (FF) 24 μg; Test type: Superiority; p = 0.006, Mixed Models Analysis; LSMean difference = 0.044, 95% CI 2-sided [0.013 to 0.076]
Statistical Analysis 9: Comparison: Formoterol Fumarate (FF) 12 μg vs Perforomist 20 μg; Test type: Superiority; p = 0.756, Mixed Models Analysis; LSMean difference = 0.005, 95% CI 2-sided [-0.026 to 0.036]
Statistical Analysis 10: Comparison: Formoterol Fumarate (FF) 24 μg vs Perforomist 20 μg; Test type: Superiority; p = 0.014, Mixed Models Analysis; LSMean difference = -0.039, 95% CI 2-sided [-0.071 to -0.008]

2. Secondary Outcome: Change From Baseline in FEV1 AUC0-6/6h at Day 1 on Treatment
Description: To assess the bronchodilation of 3 doses of formoterol fumarate (6 μg, 12 μg and 24 μg) BID administered via Pressair® compared to placebo and to open-label nebulised formoterol fumarate (20 μg and 40 μg). 6-hour serial spirometry was performed at Day 1 of each treatment period: spirometry was performed post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours and 6 hours post-dose.
Time Frame: Day 1: zero time to 6 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litre/Hour
Groups:
- Perforomist 40 μg: Randomized participants received single dose of 2 vials of Perforomist 20 μg oral nebulization solution via a jet nebulizer in the morning of Day 1 of assigned treatment period.
Arm/Group | Formoterol Fumarate 6 μg | Formoterol Fumarate (FF) 12 μg | Formoterol Fumarate (FF) 24 μg | Perforomist 20 μg | Perforomist 40 μg | Placebo (Lactose Monohydrate)
Number analyzed (Participants) | 106 | 121 | 104 | 118 | 108 | 38
Litre/Hour | 0.111 [0.077 to 0.145] | 0.148 [0.115 to 0.182] | 0.205 [0.171 to 0.239] | 0.195 [0.162 to 0.229] | 0.246 [0.212 to 0.280] | -0.019 [-0.063 to 0.025]
Statistical Analysis 1: Comparison: Formoterol Fumarate 6 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.130, 95% CI 2-sided [0.091 to 0.169]
Statistical Analysis 2: Comparison: Formoterol Fumarate (FF) 12 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.167, 95% CI 2-sided [0.128 to 0.206]
Statistical Analysis 3: Comparison: Formoterol Fumarate (FF) 24 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.224, 95% CI 2-sided [0.184 to 0.263]
Statistical Analysis 4: Comparison: Perforomist 20 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.214, 95% CI 2-sided [0.176 to 0.253]
Statistical Analysis 5: Comparison: Perforomist 40 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.265, 95% CI 2-sided [0.226 to 0.304]
Statistical Analysis 6: Comparison: Formoterol Fumarate 6 μg vs Formoterol Fumarate (FF) 12 μg; Test type: Superiority; p = 0.004, Mixed Models Analysis; LSMean difference = 0.037, 95% CI 2-sided [0.012 to 0.062]
Statistical Analysis 7: Comparison: Formoterol Fumarate 6 μg vs Formoterol Fumarate (FF) 24 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.094, 95% CI 2-sided [0.068 to 0.119]
Statistical Analysis 8: Comparison: Formoterol Fumarate 6 μg vs Perforomist 20 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.084, 95% CI 2-sided [0.059 to 0.110]
Statistical Analysis 9: Comparison: Formoterol Fumarate 6 μg vs Perforomist 40 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.135, 95% CI 2-sided [0.109 to 0.161]
Statistical Analysis 10: Comparison: Formoterol Fumarate (FF) 12 μg vs Formoterol Fumarate (FF) 24 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.057, 95% CI 2-sided [0.031 to 0.082]
Statistical Analysis 11: Comparison: Formoterol Fumarate (FF) 12 μg vs Perforomist 20 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.047, 95% CI 2-sided [0.023 to 0.071]
Statistical Analysis 12: Comparison: Formoterol Fumarate (FF) 12 μg vs Perforomist 40 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.098, 95% CI 2-sided [0.073 to 0.123]
Statistical Analysis 13: Comparison: Formoterol Fumarate (FF) 24 μg vs Perforomist 20 μg; Test type: Superiority; p = 0.469, Mixed Models Analysis; LSMean difference = -0.009, 95% CI 2-sided [-0.035 to 0.016]
Statistical Analysis 14: Comparison: Formoterol Fumarate (FF) 24 μg vs Perforomist 40 μg; Test type: Superiority; p = 0.002, Mixed Models Analysis; LSMean difference = 0.041, 95% CI 2-sided [0.015 to 0.068]
Statistical Analysis 15: Comparison: Perforomist 20 μg vs Perforomist 40 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.051, 95% CI 2-sided [0.025 to 0.076]

3. Secondary Outcome: Change From Baseline in FEV1 AUC0-6/6h at Day 7 on Treatment
Description: To assess the bronchodilation of 3 doses of formoterol fumarate (6 μg, 12 μg and 24 μg) BID administered via Pressair® compared to placebo and to open-label nebulised formoterol fumarate (20 μg). 6-hour serial spirometry was performed at Day 7 of each treatment period: spirometry was performed post-dose at 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours and 6 hours post-dose Note: Perforomist® 40 μg treatment periods lasted for 1 day only. Hence, was not included in the calculation
Time Frame: Day 7: zero time to 6 hours post-dose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litre/Hour
Arm/Group | Formoterol Fumarate 6 μg | Formoterol Fumarate (FF) 12 μg | Formoterol Fumarate (FF) 24 μg | Perforomist 20 μg | Placebo (Lactose Monohydrate)
Number analyzed (Participants) | 105 | 119 | 104 | 117 | 36
Litre/Hour | 0.166 [0.127 to 0.205] | 0.177 [0.139 to 0.215] | 0.225 [0.186 to 0.265] | 0.186 [0.147 to 0.225] | 0.007 [-0.050 to 0.064]
Statistical Analysis 1: Comparison: Formoterol Fumarate 6 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.159, 95% CI 2-sided [0.105 to 0.213]
Statistical Analysis 2: Comparison: Formoterol Fumarate (FF) 12 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.170, 95% CI 2-sided [0.116 to 0.224]
Statistical Analysis 3: Comparison: Formoterol Fumarate (FF) 24 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.219, 95% CI 2-sided [0.163 to 0.274]
Statistical Analysis 4: Comparison: Perforomist 20 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.179, 95% CI 2-sided [0.125 to 0.233]
Statistical Analysis 5: Comparison: Formoterol Fumarate 6 μg vs Formoterol Fumarate (FF) 12 μg; Test type: Superiority; p = 0.488, Mixed Models Analysis; LSMean difference = 0.011, 95% CI 2-sided [-0.020 to 0.042]
Statistical Analysis 6: Comparison: Formoterol Fumarate 6 μg vs Formoterol Fumarate (FF) 24 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 0.060, 95% CI 2-sided [0.027 to 0.092]
Statistical Analysis 7: Comparison: Formoterol Fumarate 6 μg vs Perforomist 20 μg; Test type: Superiority; p = 0.206, Mixed Models Analysis; LSMean difference = 0.020, 95% CI 2-sided [-0.011 to 0.051]
Statistical Analysis 8: Comparison: Formoterol Fumarate (FF) 12 μg vs Formoterol Fumarate (FF) 24 μg; Test type: Superiority; p = 0.004, Mixed Models Analysis; LSMean difference = 0.049, 95% CI 2-sided [0.016 to 0.081]
Statistical Analysis 9: Comparison: Formoterol Fumarate (FF) 12 μg vs Perforomist 20 μg; Test type: Superiority; p = 0.567, Mixed Models Analysis; LSMean difference = 0.009, 95% CI 2-sided [-0.022 to 0.041]
Statistical Analysis 10: Comparison: Formoterol Fumarate (FF) 24 μg vs Perforomist 20 μg; Test type: Superiority; p = 0.017, Mixed Models Analysis; LSMean difference = -0.039, 95% CI 2-sided [-0.072 to -0.007]

4. Secondary Outcome: Change From Baseline in Morning Pre-dose (Trough) FEV1 at Day 7 on Treatment
Description: To assess the bronchodilation of 3 doses of formoterol fumarate (6 μg, 12 μg and 24 μg) BID administered via Pressair® compared to placebo and to open-label nebulised formoterol fumarate (20 μg). Trough value was defined as the mean of the 2 pre-dose measurements on Day 7. If 1 of the 2 measurements was missing, the non-missing measurement was used as the trough value.
  Note: Perforomist® 40 μg treatment periods lasted for 1 day only. Hence, was not included in the calculation.
Time Frame: At baseline and Day 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Litre
Arm/Group | Formoterol Fumarate 6 μg | Formoterol Fumarate (FF) 12 μg | Formoterol Fumarate (FF) 24 μg | Perforomist 20 μg | Placebo (Lactose Monohydrate)
Number analyzed (Participants) | 105 | 119 | 104 | 117 | 36
Litre | 0.077 [0.044 to 0.109] | 0.067 [0.035 to 0.098] | 0.102 [0.069 to 0.135] | 0.061 [0.029 to 0.092] | 0.002 [-0.059 to 0.063]
Statistical Analysis 1: Comparison: Formoterol Fumarate 6 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p = 0.027, Mixed Models Analysis; LSMean difference = 0.075, 95% CI 2-sided [0.008 to 0.141]
Statistical Analysis 2: Comparison: Formoterol Fumarate (FF) 12 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p = 0.054, Mixed Models Analysis; LSMean difference = 0.065, 95% CI 2-sided [-0.001 to 0.131]
Statistical Analysis 3: Comparison: Formoterol Fumarate (FF) 24 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p = 0.004, Mixed Models Analysis; LSMean difference = 0.100, 95% CI 2-sided [0.032 to 0.168]
Statistical Analysis 4: Comparison: Perforomist 20 μg vs Placebo (Lactose Monohydrate); Test type: Superiority; p = 0.075, Mixed Models Analysis; LSMean difference = 0.059, 95% CI 2-sided [-0.006 to 0.123]
Statistical Analysis 5: Comparison: Formoterol Fumarate 6 μg vs Formoterol Fumarate (FF) 12 μg; Test type: Superiority; p = 0.615, Mixed Models Analysis; LSMean difference = -0.010, 95% CI 2-sided [-0.048 to 0.028]
Statistical Analysis 6: Comparison: Formoterol Fumarate 6 μg vs Formoterol Fumarate (FF) 24 μg; Test type: Superiority; p = 0.209, Mixed Models Analysis; LSMean difference = 0.025, 95% CI 2-sided [-0.014 to 0.065]
Statistical Analysis 7: Comparison: Formoterol Fumarate 6 μg vs Perforomist 20 μg; Test type: Superiority; p = 0.403, Mixed Models Analysis; LSMean difference = -0.016, 95% CI 2-sided [-0.053 to 0.022]
Statistical Analysis 8: Comparison: Formoterol Fumarate (FF) 12 μg vs Formoterol Fumarate (FF) 24 μg; Test type: Superiority; p = 0.074, Mixed Models Analysis; LSMean difference = 0.035, 95% CI 2-sided [-0.003 to 0.074]
Statistical Analysis 9: Comparison: Formoterol Fumarate (FF) 12 μg vs Perforomist 20 μg; Test type: Superiority; p = 0.750, Mixed Models Analysis; LSMean difference = -0.006, 95% CI 2-sided [-0.045 to 0.032]
Statistical Analysis 10: Comparison: Formoterol Fumarate (FF) 24 μg vs Perforomist 20 μg; Test type: Superiority; p = 0.035, Mixed Models Analysis; LSMean difference = -0.041, 95% CI 2-sided [-0.080 to -0.003]

ADVERSE EVENTS:
Time Frame: From the time of signature of informed consent throughout the treatment period and including the follow-up period (i.e. 2 weeks after the last IP).
Description: Adverse event: The development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition can be symptoms (e.g., nausea, chest pain), signs (e.g., tachycardia, enlarged liver) or the abnormal results of an investigation (e.g., laboratory findings, electrocardiogram)
Arm/Group | Formoterol Fumarate 6 μg | Formoterol Fumarate (FF) 12 μg | Formoterol Fumarate (FF) 24 μg | Perforomist 20 μg | Perforomist 40 μg | Placebo (Lactose Monohydrate)
All-Cause Mortality (participants affected / at risk) | 0/107 | 1/121 | 0/105 | 0/118 | 0/109 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/107 | 2/121 | 0/105 | 0/118 | 1/109 | 1/38
Other Adverse Events (participants affected / at risk) | 3/107 | 4/121 | 1/105 | 7/118 | 0/109 | 3/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Formoterol Fumarate 6 μg (N=107) | Formoterol Fumarate (FF) 12 μg (N=121) | Formoterol Fumarate (FF) 24 μg (N=105) | Perforomist 20 μg (N=118) | Perforomist 40 μg (N=109) | Placebo (Lactose Monohydrate) (N=38)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vascular stent occlusion (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Formoterol Fumarate 6 μg (N=107) | Formoterol Fumarate (FF) 12 μg (N=121) | Formoterol Fumarate (FF) 24 μg (N=105) | Perforomist 20 μg (N=118) | Perforomist 40 μg (N=109) | Placebo (Lactose Monohydrate) (N=38)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 3 | 1 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.